CLINICAL TRIAL: NCT07080424
Title: Comparison of Post-Operative Wound Healing in Fistulectomy and Fistulectomy With Marsupialization in Patients With Low Fistula in Ano
Brief Title: Comparison of Wound Healing in Fistulectomy and Fistulectomy With Marsupialization
Status: Completed | Type: Observational
Sponsor: Central Park Medical College (Other)
Responsible Party: Principal Investigator, Mirza Zeeshan Sikandar, Principal Investigator, Central Park Medical College
Other Study IDs: PHRF/2023/S23
Record Dates: First submitted 2025-07-07; First posted 2025-07-23 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Wound Healing; Fistulectomy; Fistulectomy With Marsupialization; Fistula in Ano
MeSH Terms: conditions — Rectal Fistula

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: patients undergoing Fistulectomy with Marsupialization
  Interventions: Procedure: Fistulectomy with Marsupialization
- Group 2: patients undergoing Fistulectomy only
  Interventions: Procedure: Fistulectomy

INTERVENTIONS:
Procedure: Fistulectomy with Marsupialization — Patients with fistula in ano treated with Fistulectomy with Marsupialization and were compared for wound healing with other group
  Groups: Group 1
Procedure: Fistulectomy — Patients with fistula in ano treated with Fistulectomy and were compared for wound healing with other group
  Groups: Group 2

SUMMARY:
The study was done at Central Park Medical College Lahore during January to September, 2024. Low fistula-in-ano patients were randomized into 2 groups i.e. Group A (SUR 1 fistulectomy) and Group B (170 patients in each group). The same surgical team applied all their procedures to reach spinal anesthesia. Wound infection determined after the operation was done clinically and verified by culture at 10 days of follow up. Statistical analyses based on SPSS version 26 were carried out and p < 0.05 terminated as significant.

ELIGIBILITY:
Inclusion Criteria:

Patients of either gender aged between 18-70 years presenting with fistula in-ano

Exclusion Criteria:

the patients with recurrent fistula, with anal fissures, chronic colitis and hemorrhoids

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients of either gender aged between 18-70 years presenting with fistula in-ano
Sampling Method: Non-Probability Sample
Enrollment: 340 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-10-01 (Actual)

PRIMARY OUTCOMES:
Assessment of wound healing | 6 weeks
  by employing southampton scale for assessment of wound healing scale; assessment of wound healing was done

CONTACTS AND LOCATIONS:
Locations (1):
- Central Park Teaching Hospital, Lahore, Pakistan

IPD SHARING:
Plan to Share IPD: No